CLINICAL TRIAL: NCT05068869
Title: Digital Outpatient Services - a Controlled Multicenter Study
Brief Title: Digital Outpatient Services
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Heidi Holmen, Post doctor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21/06826
Record Dates: First submitted 2021-09-19; First posted 2021-10-06 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Cancer; Interstitial Lung Disease; Long Term Pain
Keywords: Digital outpatient services; Health literacy; mHealth; eHealth; Satisfaction; Controlled trial
MeSH Terms: conditions — Epilepsy; Neoplasms; Lung Diseases, Interstitial; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dignio Digital Remote Care intervention group (Other): Participants will receive the MyDignio app for individualized follow-up for 6 months.
  Interventions: Other: Dignio Digital Remote Care intervention group
- Usual Care Control group (Other): Participants in the control group will receive follow-up at the outpatient clinic as per their needs.
  Interventions: Other: Usual Care Control group

INTERVENTIONS:
Other: Dignio Digital Remote Care intervention group — The intervention consists of Dignio Prevent (for healthcare professionals) and MyDignio (for patients). The system is CE marked and the system satisfies all regulatory requirements for privacy and information security. Various components can be added for an individualized follow-up of the patients.
  Elements of the digital outpatient service in Dignio include patient reported outcomes and other questionnaires, tasks, objective measures, reminders and information, in addition to a chat function for asynchronous contact with healthcare personnel and video consultations for real-time consultations.
  Arms: Dignio Digital Remote Care intervention group
Other: Usual Care Control group — Participants in the control group will receive follow-up at the outpatient clinic as per their needs.
  Arms: Usual Care Control group

SUMMARY:
More people are living with chronic or long-term disorders together and they live longer, which gives an increase in patients who need health services. Seen in the context of the shorter lengths of stay, and the outpatient clinics' increasing responsibility, there is a need to increase outpatient capacity without leading to more patient readmissions. Further, new services should take into account the patients capacity to benefit from the services, and their level of health literacy is crucial. By developing new services using technology, patients will be able to be followed up closely in their own home with adapted treatment and information, a closer dialogue with the health service where there is a need, and the utilization of scarce resources in the health care system can increase.

The aim of the current study is to evaluate a digital outpatient clinic, and assess any differences over time in health literacy, digital health literacy, quality of life and overall satisfaction with the outpatient services. Furthermore, the investigators will assess the intervention group's satisfaction with the digital outpatient clinic. In addition, the digital services will be tailored and revised throughout the study based on continuous feedback and iterative processes.

The current study is a pragmatic controlled multicenter study with two study arms; one control arm and one intervention arm. In total, eligible participants will be recruited from one of four centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the study centers that are cognitively able to use a digital outpatient service with no major conflicting disorders, with one of the following disorders:
* cancer
* epilepsy
* interstitial lung disease
* long-term complex pain conditions

Exclusion Criteria:

* under the age of 18
* any mental or cognitive conditions interfering with their ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Health literacy | Baseline, 3 months, and 6 months follow-up.
  The HLQ is a standardized measure of health literacy, and the investigators will apply five of the nine domains; 1 Feeling understood and supported by healthcare providers; 2 Having sufficient information to manage my health; 3 Actively managing my health; 6 Ability to actively engage with healthcare providers; and 9 Understanding health information well enough to know what to do. the HLQ is is translated and validated in Norwegian.
  (Osborne et al. 2013; Wahl et al. 2020)

SECONDARY OUTCOMES:
Change in Digital health literacy | Baseline, 3 months, and 6 months months follow-up.
  The investigators will apply the eHLQ to measure level of digital health literacy. The eHLQ contains 35 items summarized in seven domains: 1) using technology to process health information, 2) understanding of health concepts and language, 3) ability to actively engage with digital services, 4) feel safe and in control, 5) motivated to engage with digital services, 6) access to digital services that work, and 7) digital services that suit individual needs. Higher scores indicate better digital health literacy. Domains 1-5 consist of 5 items, domain 6 consists of 6 items, and domain 7 consists of 4 items.
  (Kayser et al. 2018)
Change in Health/ quality of life | Baseline, 3 months, and 6 months follow-up.
  To assess the patient reported health or quality of life the investigators will use the 12-Item Short Form Survey from the RAND Medical Outcomes Study (RAND-12) (Ware et al. 1996). The items summarizes into two scales; mental component score and Physical component score. Higher scores indicate better health, and the instruments is translated and validated in Norwegian.
Change in Perceived safety in a pandemic | Baseline, 3 months, and 6 months follow-up.
  To assess the participants self-perceived safety in the pandemic the investigators will apply the item: "How anxious are you to be infected with Covid-19 (corona)?" with responses on a 5 point Likert scale from "Not anxious" to "Very anxious" .
Change in Satisfaction with digital services | 3 months, and 6 months follow-up.
  The Service User Technology Acceptability Questionnaire (SUTAQ) is an instrument that can be used to measure user beliefs about the acceptability of digital services, and has the ability to discriminate and predict individual differences in beliefs and behaviour.
  (Hirani et al 2016; Torbjørnsen et al. 2018)

OTHER OUTCOMES:
Experiences with digital outpatient services | After 6 moths of study follow-up, the investigators will conduct the interviews
  Qualitative interviews with patients and healthcare personnel will be conducted to assess their experiences with the new services.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, PhD, Study Director — Oslo University Hospital; Heidi Holmen, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmen H, Fosse E. "I Want to Spend My Time Living"-Experiences With a Digital Outpatient Service With a Mobile App for Tailored Care Among Adults With Long-Term Health Service Needs: Qualitative Study Using Thematic Analysis. J Med Internet Res. 2026 Jan 15;28:e79155. doi: 10.2196/79155. PMID 41538795
- [Derived] Holmen H, Holm AM, Falk RS, Kilvaer TK, Ljosaa TM, Ekholdt C, Fosse E. A Digital Outpatient Service With a Mobile App for Tailored Care and Health Literacy in Adults With Long-Term Health Service Needs: Multicenter Nonrandomized Controlled Trial. J Med Internet Res. 2025 Apr 28;27:e60343. doi: 10.2196/60343. PMID 40294411
- [Derived] Holmen H, Holm AM, Kilvaer TK, Ljosa TM, Granan LP, Ekholdt C, Larsen LS, Fosse E. Digital Outpatient Services for Adults: Development of an Intervention and Protocol for a Multicenter Non-Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 10;12:e46649. doi: 10.2196/46649. PMID 37428533